CLINICAL TRIAL: NCT02405936
Title: Prospective Data Collection of Patients Undergoing Gynecologic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Other Study IDs: 2014-11-009-002
Record Dates: First submitted 2015-03-28; First posted 2015-04-01 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Disease (or Disorder); Gynecological
MeSH Terms: conditions — Disease | interventions — Gynecologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gynecologic surgery — The researchers prospectively will collect data on all patients undergoing gynecologic surgery at Kangbuk Samsung Hospital since March, 2015.

SUMMARY:
The aim of this prospective study is to collect data on patients undergoing gynecologic surgery at Kangbuk Samsung Hospital.

DETAILED DESCRIPTION:
The aim of this prospective study is to collect data on patients undergoing gynecologic surgery at Kangbuk Samsung Hospital. If patients agree to participate in this clinical trial, patient's data (such as age, body mass index, preoperative findings, laboratory findings, radiologic findings, operative findings, pathologic findings, postoperative findings) will be collected in a research database. The research database will be updated, every 6 month, to include data on patient's disease outcome and follow-up care. Although most data will be collected form the medical record, patient may agin be contacted so that researchers can collection some data if it is not in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing gynecologic surgery at Kangbuk Samsung Hospital since March, 2015

Exclusion Criteria:

* None

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing gynecologic surgery at Kangbuk Samsung Hospital since March, 2015
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-03; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prospective data collection of patients undergoing gynecologic surgery | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea